CLINICAL TRIAL: NCT05976711
Title: Gamechanger: Development of MRI Based Endovascular Procedures for Vascular Surgery
Brief Title: New MRI Techniques for Diagnosis and Treatment of Patients With Abdominal Aortic Aneurysms
Acronym: MARVY
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Brightfish (Unknown); Nano4Imaging GmbH (Industry)
Responsible Party: Principal Investigator, Associate Prof. Dr. Kak Khee Yeung, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 2008987
Record Dates: First submitted 2023-07-26; First posted 2023-08-04 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-04

CONDITIONS: Abdominal Aortic Aneurysm Without Rupture
Keywords: Abdominal Aortic Aneurysm; Magnetic Resonance Imaging; 4D flow MRI; DCE MRI
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Magnetic Resonance Imaging; Dynamic Contrast Enhanced Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Surveillance: 20 AAA patients will undergo two MRI scans with a half year interval to assess a possible correlation between MRI derived biomarkers and the clinical standard to assess aneurysm progression (maximum AAA diameter).
  Interventions: Device: Magnetic resonance imaging (with PROUD software)
- EVAR planning: 10 patients will undergo magnetic resonance angiography next to the standard of CT angiography (CTA). It is investigated whether EVAR planning is feasible based on MRA and if or how measurements between MRA and CTA differ.
  Interventions: Device: Magnetic resonance imaging (with PROUD software)
- EVAR follow-up: 30 AAA patients who underwent EVAR will be included in three groups: 10 patients with ten complication free years after EVAR or sac regression, 10 patients with endoleak type I and 10 patients with endoleak type II. It is investigated whether MRI can provide extra information for the detection of endoleaks after EVAR.
  Interventions: Device: Magnetic resonance imaging (with PROUD software)

INTERVENTIONS:
Device: Magnetic resonance imaging (with PROUD software) — Philips Ingenia 3.0T MR system with in-house developed PROUD software
  Other Names: 4D flow MRI; DCE-MRI

SUMMARY:
An abdominal aortic aneurysm (AAA) is a pathological dilatation of the aorta in the belly which can rupture leading to bleeding within the belly. To prevent rupture elective surgery can be performed. Endovascular repair (EVAR) is a surgical intervention whereby a stent is inserted into the AAA to prevent it from further growth and rupture.

Standard AAA management has several drawbacks. To start: maximum AAA diameter is used to determine upon timing of elective repair but is imprecise in predicting the risk of rupture resulting in an unmet clinical need. Secondly, EVAR outcome and complication occurrence remain unpredictable due to poor prediction ability of computed tomography (CT) and ultrasound (US) utilised in the follow-up protocol. Lastly, patients and physicians are being repeatedly exposed to cumulative radiation toxicity. All these drawbacks could be solved by trading the standard imaging modalities by magnetic resonance imaging (MRI). Within the MARVY, advanced MRI techniques are used to find out if standard imaging techniques could be replaced by MRI in three phases of the AAA management (surveillance, surgery planning and post-operative follow-up). The two most important MRI techniques that will be used are 4D flow MRI and dynamic contrast enhanced (DCE) MRI which give respectively information about the blood flow within the AAA and perfusion of the aortic wall.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with AAA
* provision of written informed consent

Inclusion Criteria for surveillance part:

* maximum AAA diameter between 3-5 cm
* not scheduled for aneurysm repair at the time of inclusion

Inclusion Criteria for planning part:

* planned for elective EVAR

Inclusion Criteria for follow-up part:

* ten complication free years after EVAR or sac regression after EVAR; or
* type I endoleak after EVAR; or
* type II endoleak after EVAR;

Exclusion Criteria:

* Supra- or pararenal AAA
* Inflammatory, infectious or mycotic AAA
* Vasculitis and connective tissue disease
* Patients that underwent open surgical repair for their AAA
* Patients with ruptured AAAs
* Patients that previously presented with allergic reactions to intravenous contrast agents

Exclusion Criteria for surveillance part:

* previous AAA repair
* severely reduced renal function
* previous allergic reactions to intravenous contrast agents

Exclusion Criteria for planning part:

* previous AAA repair

Exclusion Criteria for follow-up part:

* severely reduced renal function
* previous allergic reactions to intravenous contrast agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an AAA from the Amsterdam UMC
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Surveillance: correlation between growth rate and MRI derived parameters | 1 year
  The main study parameter for phase B1 (surveillance) is the correlation between growth rate of the AAA (determinant for the standard of care) and measured MRI parameters acquired with 4D flow MRI and DCE-MRI.
EVAR planning: correlation between morphological parameters measured based on MRA and CTA | half year
  The main study parameter for phase B2 (EVAR planning) is the difference between anatomical measurements (lengths and diameters) based on both CTA and MRA. Several quantitative anatomical measurements will be utilised to assess the feasibility of MRA for planning of EVARs.
EVAR follow up: difference in MRI parameters between patients with endoleaks and without | 1 year
  The main study parameter for phase B3 (EVAR follow-up) is the difference in MRI parameters measured post-operatively in patients with and without EVAR related complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No